CLINICAL TRIAL: NCT00005916
Title: A Randomized Phase II Study of a PSA-Based Vaccine in Patients With Localized Prostate Cancer Receiving Standard Radiotherapy
Brief Title: PSA-Based Vaccine and Radiotherapy to Treat Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000154; 00-C-0154; NCT00020228 (obsolete NCT alias)
Record Dates: First submitted 2006-06-30; First posted 2000-06-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2005-12-22

CONDITIONS: Prostate Cancer; Prostate Neoplasm
Keywords: Immunotherapy; Radiation; Immunology; Prostvac; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC

INTERVENTIONS:
Drug: rV-PSA
Drug: rF-PSA
Drug: rV-B7.1

SUMMARY:
This study will test the ability of an experimental vaccine to increase the number of tumor-fighting immune cells (lymphocytes) in patients with localized prostate cancer and prevent the disease from recurring following radiation therapy. The vaccine is intended to stimulate lymphocytes to target and attack cells containing a protein called prostate specific antigen, or PSA. It is composed of the following parts:

* rV-PSA: Vaccinia virus plus human DNA that produces PSA (prostate specific antigen)
* rV-B7.1: Vaccinia virus plus human DNA that produces B7.1 (a protein that helps guide immune cells to their targets)
* rF-PSA: Fowlpox virus plus human DNA that produces PSA
* GM-CSF: Drug that boosts the immune system.
* IL-2: Drug that boosts the immune system.

Patients 18 years of age and older with prostate cancer confined to the prostate who have received a smallpox vaccine sometime in the past and who do not have a history of allergy to eggs may be eligible for this study. Candidates are screened with a complete medical history and physical examination, blood tests, and skin tests (similar to those for allergies or tuberculosis) to assess immune function.

Participants are randomly assigned to receive one of the following three treatments: Group 1 - standard radiation therapy plus the experimental vaccine; Group 2 - standard radiation therapy without the vaccine; Group 3 - standard radiation therapy with the vaccine, but with a different dose of IL-2 from Group 1.

Patients in the vaccine groups receive injections in the arm or thigh in 28-day treatment cycles, as follows:

* GM-CSF: Days 1 through 4 of the first week
* IL-2 5: for Group 1, 5 days in the second week of each cycle; for Group 3, 14 days beginning in the second week of each cycle
* rV-PSA and rV-B7.1: Day 2 of the first cycle only
* rF-PSA (booster shots): Every 28 days, beginning day 2 of the second cycle (i.e., days 30, 58, 86, etc.)

Treatment continues for eight cycles unless serious side effects develop, PSA levels rise significantly, or the doctors feel there is no reason to continue therapy.

All patients undergo radiation therapy and possibly hormone therapy, if indicated. Blood samples are drawn once a week for the first month and then once every 4 weeks to monitor safety. After treatment ends, patients are followed with examinations and blood tests every 3 months for the first 2 years and then every 6 months until the doctors determine follow-up is no longer needed or the cancer returns.

All patients have HLA tissue typing at the beginning of the study. Those who are type HLA-A2 are asked to have additional procedures for studying the immune response that can be done only with this tissue type. This involves collecting blood samples before treatment begins, every 4 weeks during treatment, once after cycle 2, and once 4 months after the eighth vaccine. They also undergo four leukapheresis procedures for collecting white blood cells. For leukapheresis, blood is collected through a needle in an arm vein, similar to donating a unit of blood. The blood flows through a machine that separates it into its components. The white cells are removed, and the red cells, platelets and plasma are returned to the body, either through the same needle or through a needle in the other arm.

DETAILED DESCRIPTION:
This trial will evaluate the immunologic effects of a vaccination regimen in HLA-A2 positive prostate cancer patients. Eligible patients will have localized prostate cancer and be willing to undergo definitive local radiotherapy. 30 patients will be randomized in a 2:1 ratio into two cohorts (see schema below) with patients in the vaccine arm receiving vaccination before, during and after primary standard radiotherapy (external beam alone or in combination with brachytherapy). When enrollment to these two cohorts is complete, enrollment will begin with up to 19 (9-10 HLA-A2 positive) patients to a third, non-randomized vaccine cohort. This cohort C will differ from the first vaccine cohort only in the IL-2 dose and schedule. The vaccine regimen will be composed of (1) a recombinant vaccinia virus that expresses the Prostate Specific Antigen gene (rV-PSA), admixed with (2) a recombinant vaccinia virus that expresses B7.1 costimulatory molecule (rV-B7.1); followed by (3) sequential vaccinations with recombinant fowlpox virus containing the PSA gene (rF-PSA). All patients on the vaccine arms will, in addition, receive sargramostim and aldesleukin as part of their vaccination schedule.

The primary endpoint is to identify immunologic response as measured by in vitro analysis of the patients peripheral blood cells. The immune response of cohorts A and B will be analyzed at various times to determine whether a specific immune response can be affected by the vaccination as well as whether radiotherapy has an effect on that immune response. The serum PSA will be followed as a secondary endpoint.

All patients with PSA-expressing adenocarcinoma of the prostate will be evaluated for eligibility that includes a history of prior vaccinia (as vaccine against smallpox) and immunocompetence.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with histologically confirmed diagnosis of adenocarcinoma of the prostate who are candidates for definitive radiotherapy, who have not had local therapy but who agree to be treated with radiotherapy (external beam therapy alone or in combination with brachytherapy).

Patients must be HLA-A2 positive for cohorts A and B. At least 9 patients must be HLA-A2 positive in cohort C.

Zubrod (ECOG) performance 0-1.

Age greater than or equal to 18 years.

Concurrent hormonal therapy will be allowed.

Patients must have received prior vaccinia (for smallpox immunization). For patients less than 30 years of age, physician certification of prior smallpox immunization is required. For patients greater than or equal to age 30, patient recollection and appropriate vaccination-site scar is sufficient evidence. There must be no history of allergy or untoward reaction to prior vaccination with vaccinia virus.

Absolute lymphocyte count greater than or equal to 600/mm(3); platelets greater than or equal to 100,000/mm(3); hemoglobin greater than or equal to 8.0 grams/dl.

The initial urine analysis for eligibility should be less than or equal to grade 1 proteinuria, grade 0 hematuria and no abnormal sediment. Any positive protein, including trace values, should be evaluated by a 24-hour urine less than or equal to 1 gram per 24 hours. Any other abnormalities in the sediment or the presence of hematuria should be evaluated by a nephrologist for evidence of underlying renal pathology. Patients may be eligible if the underlying cause of the abnormality is determined to be non-renal.

Serum bilirubin less than or equal to 1.6 mg/dl, AST and ALT less than or equal to 4 times normal; serum creatinine less than or equal to 1.5 mg/dl or a creatinine clearance of greater than 60 ml/min.

Patients must understand and sign informed consent that explains the neoplastic nature of his disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, potential risks and toxicities, and the voluntary nature of participation.

EXCLUSION CRITERIA:

Patients should have no evidence of being immunocompromised as listed below:

They should have no reactive HIV testing;

They should not have any other diagnosis of altered immune function, autoimmune disease (autoimmune neutropenia, thrombocytopenia, or hemolytic anemia; systemic lupus erythematosus, Sjogren syndrome, or scleroderma; myasthenia gravis; Goodpasture syndrome; Addison's disease, Hashimoto's thyroiditis, or active Graves' disease).

They should not have prior radiation therapy greater than 50% of nodal groups;

They should not have had a prior splenectomy;

They should not be using glucocorticoids (including glucocorticoids for brachytherapy).

The recombinant vaccinia vaccine should not be administered if the following apply to either recipients or, for at least two weeks after vaccination, their close household contacts: Persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne or other open rashes or wound) until condition resolves; Pregnant or nursing women; Children under 5 years of age; and immunodeficient or immunosuppressed persons (by disease or therapy) , including HIV infection. Close household contacts are those who share housing or have close physical contact.

Other serious intercurrent illness. Patients with active infections requiring antibiotic treatment (including chronic suppressive therapy) are not eligible until the infection has cleared and the antibiotics have been stopped for at least three days.

History of other malignant process (excluding squamous cell or basal cell carcinoma of the skin), unless that previous tumor was treated with curative intent and the patient has been in remission for at least three years.

Patients with a history of seizures, encephalitis, or multiple sclerosis are not eligible.

Patients with known allergy to eggs are not eligible.

Patients should not have any cardiac disease, pulmonary disease, autoimmune disease, renal disease or hepatic dysfunction that may be exacerbated by IL-2.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2000-06-13; Study Completion 2005-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lechleider RJ, Arlen PM, Tsang KY, Steinberg SM, Yokokawa J, Cereda V, Camphausen K, Schlom J, Dahut WL, Gulley JL. Safety and immunologic response of a viral vaccine to prostate-specific antigen in combination with radiation therapy when metronomic-dose interleukin 2 is used as an adjuvant. Clin Cancer Res. 2008 Aug 15;14(16):5284-91. doi: 10.1158/1078-0432.CCR-07-5162. PMID 18698048
- [Background] Gulley JL, Arlen PM, Bastian A, Morin S, Marte J, Beetham P, Tsang KY, Yokokawa J, Hodge JW, Menard C, Camphausen K, Coleman CN, Sullivan F, Steinberg SM, Schlom J, Dahut W. Combining a recombinant cancer vaccine with standard definitive radiotherapy in patients with localized prostate cancer. Clin Cancer Res. 2005 May 1;11(9):3353-62. doi: 10.1158/1078-0432.CCR-04-2062. PMID 15867235
- [Background] Nesslinger NJ, Ng A, Tsang KY, Ferrara T, Schlom J, Gulley JL, Nelson BH. A viral vaccine encoding prostate-specific antigen induces antigen spreading to a common set of self-proteins in prostate cancer patients. Clin Cancer Res. 2010 Aug 1;16(15):4046-56. doi: 10.1158/1078-0432.CCR-10-0948. Epub 2010 Jun 18. PMID 20562209
- [Background] Yokokawa J, Cereda V, Remondo C, Gulley JL, Arlen PM, Schlom J, Tsang KY. Enhanced functionality of CD4+CD25(high)FoxP3+ regulatory T cells in the peripheral blood of patients with prostate cancer. Clin Cancer Res. 2008 Feb 15;14(4):1032-40. doi: 10.1158/1078-0432.CCR-07-2056. PMID 18281535